CLINICAL TRIAL: NCT00134303
Title: Double Blinded Randomised Trial Comparing Metformin Versus Placebo in NASH Patients Receiving Bariatric Surgery for Obesity
Brief Title: Trial Comparing Metformin Versus Placebo in Non Alcoholic Steatohepatitis (NASH) Patients Receiving Bariatric Surgery for Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2005/045
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- NASH (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin is used.

SUMMARY:
This is a comparison of metformin versus placebo in NASH patients receiving bariatric surgery for obesity.

DETAILED DESCRIPTION:
In patients receiving bariatric surgery, a preoperative liver biopsy will confirm the presence of NASH. Those patients with NASH (histologically defined according the Brunt's criteria) will be randomized to receive metformin (2 times 850 mg orally daily) or placebo for a time period of 1 year. A control liver biopsy will be performed after one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving bariatric surgery for obesity

Exclusion Criteria:

* Other causes of liver disease (hepatitis B virus [HBV], hepatitis C virus [HCV], primary biliary cirrhosis [PBC], etc.)
* Patients with diabetes type I
* Patients with endocrinological reasons for obesity (eg. Cushing, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2005-06; Primary Completion 2006-03-31 (Actual); Study Completion 2006-03-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with histological amelioration of NASH after a period of 1 year | 1 year

SECONDARY OUTCOMES:
Number of patients with normalisation of ALT, steatosis on ultrasound after a period of 1 year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hans Van Vlierberghe, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be